CLINICAL TRIAL: NCT01799486
Title: Telbivudine Renoprotective Effect in Patients With the HBV-related Liver Cirrhosis: a Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lin Bingliang (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Lin Bingliang, The Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Professor Bingliang Lin
Record Dates: First submitted 2013-02-19; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: HBV-related Liver Cirrhosis
Keywords: Telbivudine; renoprotective efficacy; liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Telbivudine; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Telbivudine (Experimental): Telbivudine,600mg/d,oral,100patients,2 years.
  Interventions: Drug: Telbivudine
- Adefovir (Experimental): Adefovir,10mg/d,oral,100 patients,2years.
  Interventions: Drug: Enecavir
- Enecavir (Experimental): Enecavir,0.5mg/d,oral,100 patients,2 year
  Interventions: Drug: Adefovir

INTERVENTIONS:
Drug: Telbivudine — 600 mg monotherapy supplied in film-coated tablets.
  Other Names: No.
  Arms: Telbivudine
Drug: Enecavir — 0.5 mg monotherapy supplied in tablets.
  Other Names: No.
  Arms: Adefovir
Drug: Adefovir — 10 mg monotherapy supplied in tablets.
  Other Names: No.
  Arms: Enecavir

SUMMARY:
Chronic hepatitis B virus (HBV) infection is a serious clinical problem because of its worldwide distribution and potential adverse outcome, including cirrhosis, which is a major cause of HBV related death. Studies show the use of nucleot(s)ide analogs treatment can alleviate, even reverse the progress of HBV-related cirrhosis. In cirrhosis stage, some potential factors, including endocrine disorder, renin, aldosterone, vasopressin increasing, hepatitis B virus related nephritis, hepatorenal syndrome, may cause renal damage. With the exposure of NAs, adverse reports of rhabdomyolysis, renal dysfunction, and lactic acidosis are increasing. So when choosing NAs, the potential renal function impairment should be considered.

Recently, Gane, Xiaoxi Li have separately reported that Telbivudine can improve estimate of glomerular filtration rate (eGFR) of patients with chronic hepatitis B, while eGFR of patients with Lamivudine, adefovir and entecavir have a trend of decrease, which suggested Telbivudine may have renal protective effects. This effect on patients with HBV-related liver cirrhosis has not been studied, which is not clear now.

This study is a randomized controlled study to prospectively observe Telbivudine's effect on renal function, which aims to provide evidence in antiviral treatment for the patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:Subjects eligible for enrolment in the study must meet all of the following criteria:

* eGFR in baseline less than 90 ml.min-1.1.73m2
* Aged between 18-75 years (inclusive).
* Male or female.
* Subjects with positive HBsAg for more than 6 months and anti-HBs negative regardless of HBeAg status. If eAg+, HBV DNA ≥2×104 IU/ml and <2×108 IU/ml; If eAg-, HBV DNA ≥2×103 IU/ml and <2×106 IU/ml.
* Subjects with HBV-related liver cirrhosis, including compensated cirrhosis and decompensated, but only Child-Pugh A or B. Cirrhosis was diagnosed by the evidence of a small, nodular liver, as shown by ultrasound, computerized omography (CT), and magnetic resonance (MR), with the exclusion of primary biliary cirrhosis and cirrhosis caused by schistosome.
* The ablility to understand and sign a written informed consent prior to any study related procedure and comply with the requirements of the study.

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study

* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures
* Patient is pregnant or breastfeeding.
* Subjects with non-HBV cirrhosis
* Co-infection with HAV/HCV/HDV/ HIV
* Patients who have previously been involved in a trial with telbivudine.
* Patient has received nucleoside or nucleotide drugs whether approved or investigational at any time.
* Patient has received IFN or other immunomodulatory treatment in the 6 months before Screening for this study.
* Patient has a history of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin. Patients with previous findings suggestive of possible hepatocellular carcinoma (HCC), should have the disease ruled out prior to entrance into the study.
* Patient has one or more additional known primary or secondary causes of liver disease other than CHB, including steatohepatitis，autoimmune hepatitis and so on. Gilbert's syndrome and Dubin-Johnson syndrome are not considered exclusion criteria for this study.
* History of any other acute or chronic medical condition that in the opinion of the investigator would make the patient unsuitable for inclusion into the study.
* Patient is currently abusing alcohol or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding two years.
* Patient has a medical condition that requires frequent or prolonged use of systemic corticosteroids, although inhaled corticosteroids are allowed.
* Patient has a history of clinical and laboratory evidence of chronic renal insufficiency.
* Patient has a medical condition requiring the chronic or prolonged use of potentially hepatotoxic drugs or nephrotoxic drugs.
* Patient has any other concurrent medical or social condition likely to preclude compliance with the schedule of evaluations in the protocol, or likely to confound the efficacy or safety observations of the study.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* Patient has a history of myopathy, myositis, or persistent muscle weakness.
* Kidney impairment due to non-HBV factors
* Inability to comply with study requirements as determined by the study investigator
* Patients with eGFR≤15 ml.min-1.1.73m2, who may need dialysis or renal transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Change of estimate of glomerular filtration rate (eGFR)* and Serum creatinine in week 4,12,18,24,48,72,96 in each Group. | up to 2years
  NO.

SECONDARY OUTCOMES:
Liver function change (ALB/GLB, ALT/AST, TB) in each Group | up to 2 years

OTHER OUTCOMES:
Percentage of subjects with ALT normalization rate at year 1and year 2 in each Group. | up to 2 years
The rate of complications (ascites, hepatorenal syndrome and so on) | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Bingliang, PhD, Study Chair — Department of Infectious Diseases, The Third Affiliated Hospital of Sun Yat-sen University